CLINICAL TRIAL: NCT00158236
Title: Effects of Buprenorphine/Naloxone in Non-Dependent Opioid Abusers
Brief Title: Abuse Potential of Buprenorphine and Naloxone in Non-Dependent Opioid Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08045-5; R01-08045-5; DPMC
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2006-01

CONDITIONS: Opioid-Related Disorders
Keywords: Opiate Addiction; Opiate Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination; Hydromorphone

INTERVENTIONS:
Drug: Buprenorphine
Drug: Buprenorphine and Naloxone
Drug: Hydromorphone

SUMMARY:
Buprenorphine is a medication used to treat opioid addiction, but individuals who use this drug are at risk of abusing it. A buprenorphine and naloxone combination may reduce the likelihood of buprenorphine addiction. This study will evaluate the potential for abuse of buprenorphine and a buprenorphine and naloxone combination in non-dependent opioid users.

DETAILED DESCRIPTION:
Opioid withdrawal symptoms are a major contributing factor for why opioid treatment programs often fail. Individuals with severe opioid withdrawal may experience shaking, muscle and bone pain, nausea, depression, anxiety, and drug craving. Buprenorphine, a medication that is used to treat opioid addiction, works by lessening the withdrawal symptoms. However, past research has shown that individuals who use buprenorphine are at risk for abusing the drug. Naloxone, another medication, is currently used to treat substance addiction. It is also used in combination with buprenorphine to reduce the risk of buprenorphine abuse in individuals who are physically dependent upon opioids. The purpose of this study is to compare the abuse potential of buprenorphine versus a buprenorphine and naloxone combination in non-dependent opioid users.

This 7-week study will enroll non-dependent opioid users. Participants will take part in two medication challenge sessions per week. At each challenge session, participants will be randomly assigned to receive varying doses of either buprenorphine; a buprenorphine and naloxone combination; hydromorphone, which is a medication used to treat moderate to severe pain; or placebo. Buprenorphine and naloxone will be administered as tablets that are dissolved under the tongue. Hydromorphone will be injected. During the challenge sessions, participants will complete performance tasks to measure psychomotor and cognitive functioning. Questionnaires and self-reports will be completed to assess medication effects. Heart rate and blood pressure will be monitored throughout all sessions, and a specialized camera will be used to assess pupillary response of the eyes.

ELIGIBILITY:
Inclusion Criteria:

* Current opioid abuse
* Not physically dependent on opioids

Exclusion Criteria:

* Significant medical or psychiatric illness (e.g., insulin-dependent diabetes or schizophrenia)
* Seeking substance abuse treatment (will be assisted with referrals to community-based treatment programs)
* Pregnant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7
Dates: Start 1997-01; Study Completion 1998-03

PRIMARY OUTCOMES:
Opioid agonist effects (measured by Visual Analog Scale and Adjective Rating Scale during the medication challenge sessions)
Physiological effects (measured by pulse oximeter, blood pressure, heart rate, and pupillary camera during the medication challenge sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States

REFERENCES:
- [Result] Strain EC, Stoller K, Walsh SL, Bigelow GE. Effects of buprenorphine versus buprenorphine/naloxone tablets in non-dependent opioid abusers. Psychopharmacology (Berl). 2000 Mar;148(4):374-83. doi: 10.1007/s002130050066. PMID 10928310